CLINICAL TRIAL: NCT01702116
Title: Multicenter Randomized Controlled Trial, Extralevator Versus Standard Abdominoperineal Resection For Rectal Adenocarcinoma
Brief Title: Extralevator Versus Standard Abdominoperineal Resection For Rectal Adenocarcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Roberto Bergamaschi, Professor and Chief, Colon and Rectal Surgery, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APR2011
Record Dates: First submitted 2011-08-11; First posted 2012-10-05 (Estimated); Last update posted 2013-04-25 (Estimated); Status verified 2013-04

CONDITIONS: Rectal Adenocarcinoma
Keywords: rectal adenocarcinoma; Standard APR; Extralevator APR
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- extralevator APR (Experimental): This is a modified and more extensive procedure that is used to remove the levator muscle en bloc with the anal canal and the mesorectum, creating a more "cylindrical" specimen, so that the amount of tissue removed around the tumor will be larger, thereby reducing the probability that the CRM will be positive.
  Interventions: Procedure: extralevator APR
- standard APR (Active Comparator): conventional abdominoperineal resection (APR)
  Interventions: Procedure: APR

INTERVENTIONS:
Procedure: extralevator APR — Extralevator Abdominoperineal Resection For Rectal Adenocarcinoma. The aim of this modified and more extensive procedure is to remove the levator muscle en bloc with the anal canal and the mesorectum, creating a more "cylindrical" specimen, so that the amount of tissue removed around the tumor will be larger, thereby reducing the probability that the CRM will be positive.
  Arms: extralevator APR
Procedure: APR — standard Abdominoperineal Resection For Rectal Adenocarcinoma
  Arms: standard APR

SUMMARY:
This is a study that compares two types of surgery for rectal cancer. There are two procedures that can be used during this surgery, conventional abdominal resection (APR) and extended (or extralevator) APR. The investigators are doing this research to see whether the extralevator APR increases the likelihood that the edge of the tissue that is removed will be more likely to be free from cancer cells compared with the conventional APR surgery. At this time there is no evidence that one type of procedure is better at this than the other. The objective of this research is to determine whether extralevator APR is more likely to have clean margins (free of cancer) compared to the standard APR surgery.

ELIGIBILITY:
Inclusion Criteria:

* Resectable, histologically proven primary adenocarcinoma of the low rectum with internal and/or external sphincter muscle involvement. Staged as follows prior to neoadjuvant chemoradiation:
* Stage T3 or T4 at MRI
* N0-2 at MRI
* M0 at CT scan
* Patient must undergo long term neoadjuvant chemoradiation: 20 fractions of radiation over ≥5 weeks: total of 50-60 Gy, and chemotherapeutic agents

Exclusion Criteria:

* Squamous cell carcinoma
* Adenocarcinoma Stage T1-2, any N
* T4 with one of the following:

with pelvic side wall involvement requiring sacrectomy requiring prostatectomy (partial or total) Distant metastasis (M1) Unresectable primary rectal cancer or Inability to complete R0 resection. Recurrent rectal cancer Previous pelvic malignancy Inability to sign informed consent Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2011-07; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
measurement of circumferential resection margin | 0-10 minutes post surgery
  Measurement in millimeters (mm) of the circumferential resection margin.

SECONDARY OUTCOMES:
operative time | 4-6 hours
  operative time from skin incision to skin closure
hospital stay | from beginning of surgery through discharge, usually 4-5 days
  duration of hospital stay (defined as from beginning of surgery to time of discharge, measured in hours)
estimated blood loss | 4-6 hours
  estimated blood loss (ml) recorded by the anesthesiologist (not by the surgeon)

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Bergamaschi, MD, PhD, Principal Investigator — Stony Brook University Medical Center
Locations (3):
- United States (3):
  - State University Hospital Medical Center, Stony Brook, New York
  - Stony Broook University Medical Center, Stony Brook, New York
  - Stony Brook University Medical Center, Stony Brook, New York

REFERENCES:
- [Derived] Bianco F, Romano G, Tsarkov P, Stanojevic G, Shroyer K, Giuratrabocchetta S, Bergamaschi R; International Rectal Cancer Study Group. Extralevator with vs nonextralevator abdominoperineal excision for rectal cancer: the RELAPe randomized controlled trial. Colorectal Dis. 2017 Feb;19(2):148-157. doi: 10.1111/codi.13436. PMID 27369739